CLINICAL TRIAL: NCT03159897
Title: A Randomized, Open-label, Multicenter, Phase III, 2-arm Study Comparing Efficacy and Tolerability of the Intensified Variant 'Dose-dense/Dose-intense ABVD' (ABVD DD-DI) With an Interim PET Response-adapted ABVD Program as Upfront Therapy in Advanced-stage Classical Hodgkin Lymphoma (HL).
Brief Title: FIL Study on ABVD DD-DI as Upfront Therapy in HL.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL-Rouge
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Hodgkin Lymphoma
Keywords: advanced stage (IIB-IV); ABVD DD-DI; PET
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Intervention Model Description: The study aims to compare the efficacy of two alternative ABVD-based strategies, the first one (Comparator arm) based on a PET-2-adaptation, the second (Experimental arm) relying on a straight dose- and time-intensified schedule, devoid of any PET-adaptation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparator arm (Experimental): Patients will receive 2 courses of standard ABVD (ABVD-28, d1, d15, cycles of 28 days) and then proceed to interim PET/CT evaluation. Those with a PET-2-negative scan (score 1-3 on 5PS) will continue with additional 4 ABVD courses while those with a PET-2-positive (score 4-5) scan will be diverted towards an intensification phase with either escalated BEACOPP or HDT plus ASCR, according to the preference of the centre. Upon completion of treatment, patients will be categorized for response (Lugano2014) by comparing actual PET/CT imaging with baseline, whether 6 ABVD cycles or ABVDx2 + intensification phase with BEACOPP or HDT/ASCR. A salvage rescue program will be planned for patients with Stable (<PR) or Progressive Disease. ISRT 30 Gy will be delivered to complete responders (5PS score 1-2-3) on the initial bulky site(s), to focal rests in case of CR scoring 3 on 5PS with a residual size ≥ 2.5 cm and to focal rests uptakes in the event of PR scoring 4 or 5, whichever is the size.
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine
- Experimental arm (Experimental): Dose-dense and dose-intense ABVD regimen (ABVD DD-DI: intercycle 21 days, d1, d11; doxorubicin 35 mg/m2 DD 1 and 11) is given in cycles 1 to 4 and dose-dense ABVD (ABVD DD: intercycle 21 days, D1 and D11; conventional doxorubicin dose, e.g. 25 mg/m2 DD 1 and 11) is given as cycles 5 and 6). The treatment is not PET-adapted, and only patients with no response or progressive disease at interim FDG-PET as defined by the Lugano Classification (e.g., score 4 or 5 on 5PS with no significant change or with increased uptake matched with baseline and/or new FDG-avid foci consistent with lymphoma) will be diverted to salvage therapy. ISRT 30 Gy will be delivered to responder patients (DS=3), on focal PET-positive rests with a residual size ≥ 2.5 cm and on patients in PR with uptake scoring 4 or 5, whichever is the size.
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Doxorubicin — Comparator arm: cycle 1-2 (and eventually 3-6): 25 mg/m2 i.v. days 1,15. Experimental arm: Cycles 1 to 4: 35 mg/m2 i.v. days 1,11. Cycles 5 and 6: 25 mg/m2 i.v. days 1,11.
Drug: Bleomycin — Bleomicina Comparator arm: cycle 1-2 (and eventually 3-6): 10,000 units/m2 i.v. days 1,15. Experimental arm: cycles 1 to 4: 10,000 units/m2 i.v. days 1,11. Cycles 5 and 6: 10,000 units/m2 i.v. days 1,11.
Drug: Vinblastine — Vinblastina Comparator arm: cycle 1-2 (and eventually 3-6): 6 mg/m2 i.v. days 1,15. Experimental arm: cycles 1 to 4: 6 mg/m2 i.v. days 1,11. Cycles 5 and 6: 6 mg/m2 i.v. days 1,11.
Drug: Dacarbazine — Dacarbazina Comparator arm: cycle 1-2 (and eventually 3-6): 375 mg/m2 i.v. days 1,15. Experimental arm: cycles 1 to 4: 375 mg/m2 i.v. days 1,11. Cycles 5 and 6: 375 mg/m2 i.v. days 1,11.

SUMMARY:
The FIL-Rouge is a randomized, open-label, multicenter, phase III, 2-arm study. The primary objective is to compare efficacy and tolerability of the intensified variant 'dose-dense/dose-intense ABVD' (ABVD DD-DI) with an interim PET response-adapted ABVD program as upfront therapy in advanced-stage classical Hodgkin Lymphoma (HL).

DETAILED DESCRIPTION:
The study is devoted to patients affected with advanced stage (IIB-IV) Hodgkin Lymphoma.

The study aims to compare the efficacy of two alternative ABVD-based strategies, the first one (Comparator arm) based on a PET-2-adaptation, the second (Experimental arm) relying on a straight dose- and time-intensified schedule, devoid of any PET-adaptation.

In the Comparator arm, the patients will receive two courses of standard ABVD (ABVD-28). Those with a PET-2 negative scan (Deauville Score 1-3) will proceed with additional 4 ABVD courses while those with a PET-2-positive scan (Deauville score 4-5) will be diverted towards a deferred intensification with either escalated BEACOPP or HDT plus ASCR , according to the preference of the Center.

In the Experimental arm, patients are treated with three cycles of a dose-dense/dose-intense ABVD (ABVD DD-DI) [e.g. a modified ABVD including the single escalation of doxorubicin to 35 mg/m2 (70 mg/m2 per cycle) and a three-weekly recycle time for all drugs (e.g. administration of all 4 drugs at days 1 and 11 of each cycle)]. Those with a progressive disease or non-responder patients according to PET/CT imaging at interim evaluation (after cycle 3) as categorized with Lugano 2014 Classification will be diverted to salvage strategies. The other patients will receive one additional course of ABVD DD-DI followed by two courses of dose-dense three-weekly ABVD (ABVD DD) (e.g. administration of all four drugs at days 1 and 11 of each cycle at the conventional doses, including doxorubicin at 25 mg/m2).

In both treatment arms 30 Gy Involved Site Radiotherapy (ISRT) is scheduled for those patients PET-negative (DS=3) with residual tumor rests ≥ 2.5 cm and for PET-positive patients in PR (DS= 4 or 5) regardless of the size of the rests. The single reference dose is 2.0 Gy daily and fractionation is five times per week.

Only in the Comparator arm the patients in CR (final score 1-3 according to 5PS by central review panel decision) will receive adjuvant ISRT at the initial bulky site(s) for a total reference dose of 30 Gy in single daily fractions of 2.0 Gy, five times weekly.

Blinded independent central reviewing for PET imaging will supervise response categorization at interim and final PET/CT evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical HL
* Previously untreated disease
* Age 18-60 years
* Ann Arbor stage IIB with extranodal involvement and/or mediastinal bulk, III and IV (Appendix A)
* At least one target PET-avid bidimensionally assessable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2 (Appendix B)
* Adequate organ and marrow function as defined below: absolute neutrophil count >1,0 x109/L, platelets >75 x109/L
* Total bilirubin <2 mg/dl without a pattern consistent with Gilbert's syndrome
* Aspartate Transaminase and Alanine Transaminase (AST/ALT) <3 X institutional Upper Limits of Normality (ULN)
* Creatinine within normal institutional limits or creatinine clearance >50 mL/min/1.72 m2 (Appendix C)
* Females of childbearing must have a negative pregnancy test at medical supervision even if had been using effective contraception
* Life expectancy > 6 months
* Able to adhere to the study visit schedule and other protocol requirements
* Sign (or their legally acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Access to PET-CT scans facilities qualified by FIL

Exclusion Criteria:

* Nodular Lymphocyte Predominant HL
* Ann Arbor stage IIB without extranodal involvement and/or mediastinal bulky
* Prior chemotherapy or radiation therapy
* Pregnant or lactating females
* Known hypertension (as defined by the updated Guidelines [76]), cardiac arrhythmia, conduction abnormalities, ischemic cardiopathy, left ventricular hypertrophy or left ventricular ejection fraction (LVEF) ≤50% at echocardiography.
* Abnormal QTc interval prolonged (>450 msec in males; >470 msec in women)
* Diffusion lung capacity for CO (DLCO) and/or forced expiratory volume in the 1st second (FEV1) tests <50% of predicted not related to impaired respiratory capacity due to airway compression by mediastinal masses or parenchymal lymphoma
* Known cerebral or meningeal disease (HL or any other etiology)
* Prior history of malignancies unless the patient has been free of the disease for five years. Exceptions include the following: basal cells carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast and prostate cancer with TNM stage of T1a or T1b
* Uncontrolled infectious disease
* Human immunodeficiency virus (HIV) positivity or active infectious A, B or C hepatitis. HBsAg-negative patients with anti-HBc antibody and can be enrolled provided that Hepatitis B Virus (HBV)-DNA are negative and that antiviral treatment with nucleos(t)ide analogs is provided
* Uncompensated diabetes
* Refusal of adequate contraception
* Any medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 3 years
  PFS is defined as the interval elapsing from randomization until lymphoma progression or death as a result of any cause.

SECONDARY OUTCOMES:
Complete remission rate (CR rate) | 2 months and 6 months
  CR rate is defined as the proportion of patients achieving a CR after 2 months of chemotherapy (interim) and at the end of treatment
PET/CT response rate | after 2 months of chemotherapy
  PET/CT response rate
Event Free Survival (EFS) | 3 years
  EFS will be measured from the time from entry onto a study to any treatment failure including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of new treatment lacking documented progression, or death)
Disease free survival (DFS) | 3 years
  DFS will be measured from the time of occurrence of disease-free state or attainment of a CR to disease recurrence or death as a result of lymphoma or acute toxicity of treatment
Overall survival (OS) | 3 years
  OS is defined as the time from entry onto the clinical trial until death as a result of any cause
Toxicity | 6 months for acute toxicity and 5 years for late toxicity
  Acute severe toxicity, acute and delayed pulmonary toxicity, acute and delayed cardiac toxicity. Late toxicity and second malignancies.
  The severity of the toxicities will be classified according to definitions of Common Terminology Criteria for Adverse Event (CTCAE) version 4.3. It will be determined by the incidence of severe, life- threatening (CTCAE grade 3, 4 and 5) and/or serious adverse events (Infusion-related reactions).
Quality of life (QoL) | 36 months
  QoL will be measured at the baseline, the end of therapy and during follow-up through the EORTC QLQ-C30 questionnaire
Cost-effectiveness analyses | 36 months
  Cost-effectiveness analyses. ICER will be calculated by dividing the difference in mean total costs arms by the difference in the mean effects. The ICER will be calculated for the principal clinical effect measures of the trial. (i.e. PFS) and for QALYs. QALYs will be calculated multiplying the amount of time a patient spent in a particular health state by the utilities estimated using the EQ-5D questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pinto, MD, Principal Investigator — Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale - Napoli
Locations (46):
- Italy (46):
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua, Padova
  - Ospedale delle Croci - Ematologia, Ravenna, Ravenna
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C. Ematologia, Alessandria
  - Università Politecnica delle Marche, Clinica di Ematologia, Ancona
  - Ospedale C.e G. Mazzoni -U.O.C. di Ematologia, Ascoli Piceno
  - Azienda Ospedaliera S.Giuseppe Moscati -S.C. Ematologia e Trapianto emopoietico, Avellino
  - Centro Riferimento Oncologico - S.O.C. Oncologia Medica A, Aviano
  - AOU Policlinico Consorziale - U.O. Ematologia con Trapianto, Bari
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Ospedale "Monsignor Raffaele Dimiccoli" - Ematologia, Barletta
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Antonio Perrino - Ematologia, Brindisi
  - Fondazione del Piemonte per l'Oncologia - IRCCS - Ematologia, Candiolo
  - AORN S.Anna e S. Sebastiano - Oncoematologia, Caserta
  - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto
  - ASST Cremona - Ematologia e CRTO, Cremona
  - Ospedali Riuniti del Canavese, Ivrea
  - Ospedale Vito Fazzi - Ematologia, Lecce
  - Ospedale Madonna delle Grazie - Ematologia, Matera
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Ematologia, Meldola
  - Azienda Ospedali Riuniti Papardo-Piemonte - S.C. Ematologia, Messina
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - USLL13 - Dipartimento di Scienze Mediche UOC di Oncologia ed Ematologia Oncologica, Mirano
  - Azienda Ospedaliero-Universitaria Policlinico di Modena - Ematologia, Modena
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale - Ematologia Oncologica, Napoli
  - Presidio ospedaliero "A. TORTORA", Pagani
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - AOU di Parma - UO Ematologia e CTMO, Parma
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - AO di Perugia - Ematologia, Perugia
  - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - A.O.R. "San Carlo" - U.O. Ematologia, Potenza
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova - IRCCS c/o CORE (II piano), Reggio Emilia
  - Ospedale degli Infermi di Rimini, Rimini
  - IRCCS-Centro di riferimento oncologico - UO di ematologia e Trapianto Cellule Staminali, Rionero in Vulture
  - Policlinico Umberto I - Università "La Sapienza" - Istituto Ematologia -Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Policlinico Universitario Campus Bio-Medico - "Area Ematologia Trapianto Cellule Staminali Medicina Trasfusionale e Terapia cellulare", Roma
  - Università Cattolica S. Cuore - Ematologia, Roma
  - Istituto Clinico Humanitas - U.O. Ematologia, Rozzano (MI)
  - Ematologia e Trapianti A.O. San Giovanni di Dio e Ruggi D'Aragona - U.O. Ematologia, Salerno
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo
  - Univ. Perugia Sede Terni - Oncoematologia, Terni
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino - S.C.Ematologia, Torino
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase

IPD SHARING:
Plan to Share IPD: No